CLINICAL TRIAL: NCT06933004
Title: Long-term Clinical Follow-up Analysis of Patients With Lumbar Disease.
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202402029DIND
Record Dates: First submitted 2025-04-10; First posted 2025-04-17 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-03

CONDITIONS: Lumbar Disease
MeSH Terms: conditions — Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Group
  Interventions: Device: Posterior Spinal Fixation System

INTERVENTIONS:
Device: Posterior Spinal Fixation System — Using spine implants SmartMIS Spinal Fixation System or ASA Spinal Fixation System.

SUMMARY:
This study is a long-term follow-up of postoperative clinical outcomes in patients with lumbar spine disorders, monitoring spine implants SmartMIS Spinal Fixation System and ASA Spinal Fixation System.

Patients will be selected based on inclusion and exclusion criteria. The informed consent process will be initiated by the physician. A questionnaire-based survey will be conducted, which includes the Visual Analog Scale (VAS), Oswestry Disability Index (ODI), and Fusion Rate. Subjects will complete the same questionnaire assessments preoperatively and at 6 ± 3 months, 12 ± 3 months, and 24 ± 3 months postoperatively.

The total number of subjects to be enrolled is 120. The total duration of the study is expected to be 4 years.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 20 and 80 years.
2. Patients with lumbar spine disorders requiring surgical treatment.
3. Able to understand the study content after explanation, capable of expressing their experiences, and willing to sign the written informed consent form.

Exclusion Criteria:

1. Individuals with impaired decision-making capacity or from vulnerable populations.
2. Individuals who are unable or unwilling to return for follow-up assessments.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: National Taiwan University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | Preoperatively and at 6 ± 3 months, 12 ± 3 months, and 24 ± 3 months postoperatively.

SECONDARY OUTCOMES:
Oswestry Disability Index (ODI) | Preoperatively and at 6 ± 3 months, 12 ± 3 months, and 24 ± 3 months postoperatively.
Fusion Rate | Preoperatively and at 6 ± 3 months, 12 ± 3 months, and 24 ± 3 months postoperatively.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No